CLINICAL TRIAL: NCT06357949
Title: The Effectiveness of High-intensity Laser Therapy on Plantar Flexor Muscle Spasticity in Stroke
Brief Title: The Effectiveness of High-intensity Laser Therapy on Plantar Flexor Muscle Spasticity in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Atan, MD, Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-3615
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity laser therapy group (Active Comparator): High-intensity laser will be applied continuously to the gastrocnemius muscle for a total of 10 minutes with an energy density of 100 j/cm2, totaling 2500 j.
  Interventions: Device: High-intensity laser
- Sham group (Sham Comparator): The same procedure will be followed, but sham laser will be applied at 0 j/cm2 for 10 minutes.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: High-intensity laser — All patients will receive a rehabilitation program consisting of stretching, strengthening, balance, and walking exercises targeting the lower extremities for 45 minutes, 5 days a week, for 6 weeks. Walking training will initially begin on level ground and gradually progress to different levels and surfaces.
  High-intensity laser will be applied continuously in biostimulation mode 3 days a week, once a day, for a total of 9 sessions over 3 weeks
  Arms: High-intensity laser therapy group
Device: Sham laser — The same procedure will be followed, but sham laser will be applied at 0 j/cm2 for 10 minutes.
  Arms: Sham group

SUMMARY:
The aim of this study is to investigate the effectiveness of high-intensity laser therapy for treating plantar flexor muscle spasticity in subacute and chronic stroke patients, focusing on its impact on spasticity, joint range of motion, pain, muscle thickness, functional ambulation, and quality of life.

DETAILED DESCRIPTION:
Post-stroke lower limb spasticity disrupts balance and walking, often resulting in decreased walking speed, increased wheelchair use, and the need for caregiver assistance. Various approaches are utilized in spasticity management, including physical therapy, splinting, oral medications, chemical neurolysis, and surgical interventions. Laser therapy is a non-invasive, painless modality used in physiotherapy units, with a low incidence of side effects. Laser therapy has been shown to reduce muscle fatigue and increase peak torque (muscle strength) when applied before exercise. The use of high-intensity laser therapy in physiotherapy protocols has become increasingly common in recent years. Studies suggest that it enhances healing in tendons and ligaments, prevents fibrosis development, increases local blood flow and tissue regeneration, and reduces edema and pain. The aim of this study is to investigate the effectiveness of high-intensity laser therapy for treating plantar flexor muscle spasticity in subacute and chronic stroke patients, focusing on its impact on spasticity, joint range of motion, pain, muscle thickness, functional ambulation, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 and ≤ 75 years
* Patients experiencing their first stroke (onset > 3 months)
* Patients with ankle plantar flexor muscle spasticity with a Modified Ashworth Scale (MAS) score ≥ 1 and < 4
* Lower extremity Brunnstrom staging ≥ 3
* Patients describing pain complaints in the affected leg as VAS > 3.
* Patients who can stand independently or with supervision for at least 2 minutes for measurements taken while standing
* Patients who can walk independently or with/without assistive devices for at least 10 meters for measurements taken while walking
* Patients with cognitive abilities sufficient to understand the study instructions (Mini-Mental State Examination score > 23)
* Patients with stable medical and psychological conditions
* Patients willing to participate in the study

Exclusion Criteria:

* Patients with severe cardiovascular or musculoskeletal problems that impair walking (e.g., fixed ankle contracture)
* Patients who have been treated for spasticity with botulinum toxin, phenol, or alcohol injections in the past 6 months
* Patients who have undergone antispastic surgery in the treatment area in the past 6 months
* Patients with recent changes in oral antispastic medication use in the past 6 months
* Patients with acute inflammation or active infection in the treatment area
* Patients with a history of ankle joint contracture, fracture, neoplasm, vascular disease, etc.
* Patients with other neurological (Parkinson's disease, epilepsy, meningitis, cerebellar disease, vertigo, dizziness, polyneuropathy, etc.) or musculoskeletal (severe back pain, knee problems) diseases that could affect balance performance other than stroke
* Patients with severe vision, hearing, and language problems
* Patients who do not consent to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
10-Meter Walk Test | Baseline- 3 - 6 weeks(follow up)
  Test to measure patients&#39; functional ambulation skills.

SECONDARY OUTCOMES:
Modified Ashworth Scale | Baseline- 3 - 6 weeks(follow up)
  Evaluation of plantar flexor muscle spasticity using the Modified Ashworth Scale (MAS). The original Ashworth scale was a 5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension.
Joint Range of Motion (ROM) Measurement | Baseline- 3 - 6 weeks(follow up)
  Passive measurement of ankle joint range of motion (ROM) with a goniometer
Ultrasonography | Baseline- 3 - 6 weeks(follow up)
  Sonographic measurement of medial gastrocnemius muscle thickness
Timed Up and Go test | Baseline- 3 - 6 weeks(follow up)
  To determine fall risk and measure the progress of balance, sit to stand and walking
Stroke Specific Quality of Life Scale | Baseline- 3 - 6 weeks(follow up)
  It is a patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke. Scores range from 49-245.
  Higher scores indicate better functioning.
Visual analogue scale for pain (VAS- pain) | Baseline- 3 - 6 weeks(follow up)
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Atan, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital; Yunus Emre Bildik, Study Director — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoldas Aslan S, Kutlay S, Dusunceli Atman E, Elhan AH, Gok H, Kucukdeveci AA. Does extracorporeal shock wave therapy decrease spasticity of ankle plantar flexor muscles in patients with stroke: A randomized controlled trial. Clin Rehabil. 2021 Oct;35(10):1442-1453. doi: 10.1177/02692155211011320. Epub 2021 Apr 28. PMID 33906450
- [Background] Tomazoni SS, Machado CDSM, De Marchi T, Casalechi HL, Bjordal JM, de Carvalho PTC, Leal-Junior ECP. Infrared Low-Level Laser Therapy (Photobiomodulation Therapy) before Intense Progressive Running Test of High-Level Soccer Players: Effects on Functional, Muscle Damage, Inflammatory, and Oxidative Stress Markers-A Randomized Controlled Trial. Oxid Med Cell Longev. 2019 Nov 16;2019:6239058. doi: 10.1155/2019/6239058. eCollection 2019. PMID 31827687
- [Background] Pekyavas NO, Baltaci G. Short-term effects of high-intensity laser therapy, manual therapy, and Kinesio taping in patients with subacromial impingement syndrome. Lasers Med Sci. 2016 Aug;31(6):1133-41. doi: 10.1007/s10103-016-1963-2. Epub 2016 May 25. PMID 27220527